CLINICAL TRIAL: NCT04433767
Title: Nicotinic Modulation of the Cognitive Control System in Late-life Depression
Brief Title: Depressed Mood Improvement Through Nicotine Dosing 2
Acronym: DepMIND2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Warren Taylor, Professor of Psychiatry, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200457
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Depressive Disorder
Keywords: geriatrics; aging; elderly; cognition; memory; nicotine transdermal patch; depression
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transdermal Nicotine Patch (Experimental): Participants will wear open label transdermal nicotine patch daily for 12-15 weeks. They will apply study patch each morning and remove at bedtime. Dosage will begin at 3.5mg patch / day, increasing to a possible maximum of 21mg patch / day.
  Interventions: Drug: Transdermal Nicotine patch

INTERVENTIONS:
Drug: Transdermal Nicotine patch — Participants will begin a 12- week open label trial of transdermal nicotine patch during the day and remove it at night (16 hours). Dose titration starting at 3.5 mg patch/daily to maximum of 21mg patch/daily.
  After week 12 , dose will be slowly tapered over 3 weeks.
  Other Names: Nicoderm CQ; Nicotrol

SUMMARY:
Deficits in cognitive control are core features of late-life depression, contributing both to emotion dysregulation and problems with inhibiting irrelevant information, conflict detection, and working memory. Clinically characterized as executive dysfunction, these deficits are associated with poor response to antidepressants and higher levels of disability. Improvement of cognitive control network (CCN) dysfunction may benefit both mood and cognitive performance, however no current pharmacotherapy improves CCN deficits in LLD. Supported by pilot data, Investigators propose that nicotine acetylcholine receptor agonists enhance CCN function and resultantly improve mood and cognitive performance in late-life depression. The objective of this initial R61-phase trial is to first determine whether transdermal nicotine enhances CCN neural activity in an exposure-dependent fashion during an emotional response inhibition task (the emotional Stroop task). Investigator's approach for the R61 phase is to examine in 36 older adults with Major Depressive Disorder whether transdermal nicotine patches enhance CCN activity over 12 weeks as measured during fMRI with the emotional Stroop task while measuring nicotine and nicotine metabolite levels. Transdermal nicotine has a mechanism of action that is distinct from current antidepressants, potentially making it a potentially important antidepressant augmentation agent. If hypotheses are correct, as patches are commercially available, this approach could be rapidly moved into definitive studies and may have applicability to other psychiatric disorders characterized by CCN dysfunction.

DETAILED DESCRIPTION:
Late-life depression (LLD) is characterized both by affective symptoms and broad cognitive deficits. The co-occurrence of cognitive deficits in LLD, particularly executive dysfunction, is a clinically relevant phenotype characterized by significant disability and poor antidepressant response. Cognitive deficits can persist even with successful antidepressant treatment and increase the risk of depression relapse. Despite the clinical importance of cognitive deficits in LLD, there are no established treatments that specifically target cognition in this population. This is particularly important, as the cognitive deficits appear to directly contribute to disability and poor antidepressant treatment outcomes. The lack of clear pharmacologic targets and therapies aimed at improving cognitive deficits in depression is a substantial deficiency in current therapeutics.

Modulation of the cholinergic system by nicotinic receptor stimulation may improve both mood and cognition in depressed elders. Clinically, transdermal nicotine improves mood in smokers and a placebo-controlled pilot trial in nonsmoking adults found that transdermal nicotine significantly improved mood. As observed in smokers, nicotine's effect to increase cognitive control network activity while reducing default mode network activity will reduce depression's characteristic bias to negatively valenced stimuli and decrease rumination. Supporting this theory, nicotinic receptor activity stimulates serotonin release and protects against worsening mood with tryptophan depletion.

The Depressed Mind 2 Study examines whether enhancement of CCN function by nicotinic acetylcholine receptor agonists will improve mood and cognitive symptoms in LLD. This is supported by pilot data demonstrating that open-label administration of transdermal nicotine (TDN) patches safely improved depression severity. The investigators also observed trends suggesting that TDN may provide benefit for cognitive performance, specifically in domains of episodic memory, working memory, and attention. In other pilot data using an emotional Stroop task, TDN reduces the differences in functional magnetic resonance imaging (fMRI) activation in the cognitive control network (CCN) between Stroop conditions. Importantly, this activation change was associated with a corresponding reduction in depression severity. Based on these data, investigators hypothesize that nicotinic receptor agonists enhance CCN function in LLD and in turn this may improve depressive symptoms.

Thirty-six participants will be enrolled to test for target engagement, defined as TDN exposure dependent effect in CCN activation. Based on pilot data, the study will test for enhancement of CCN function by examining the Stroop fMRI response, or the reduction in CCN activation between incongruent and congruent conditions of the emotional Stroop task during fMRI. Investigators will assess the effects of variability in nicotine exposure on target engagement by measuring nicotine blood levels in conjunction with repeat MRI.

Primary aim: To test CCN engagement over 12 weeks of Open labeled Transdermal Nicotine(TDN).

Hypothesis1A(Target Engagement): TDN will enhance CCN function, measured as a reduction in the middle or superior frontal gyri (M/SFG) Stroop functional MRI response (the activation difference between incongruent and congruent conditions of the emotional Stroop task). 60% or more of subjects will exhibit a M/SFG z-score reduction of 0.5 or greater.

Hypothesis1B (Exposure): Higher nicotine exposure measured by patch dose or nicotine metabolite levels will be associated with a greater reduction in the M/SFG Stroop fMRI response.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 60 years;
2. Diagnosis of major depressive disorder, single or recurrent episode (DSM5);
3. On a stable therapeutic dose of an allowed selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) for at least 8 weeks;
4. Severity: Montgomery-Asberg Depression Rating Scale (MADRS) score ≥ 15;
5. Cognition: Mini-Mental State Examination (MMSE) score ≥ 24;
6. Fluent in English

Exclusion Criteria:

1. Other Axis I psychiatric disorders, except for generalized anxiety disorder (GAD) symptoms occurring in a depressive episode;
2. Use of other medications for depression, e.g., bupropion or augmenting agents, although short-acting sedatives are allowed (see below);
3. Any use of tobacco or nicotine in the last year;
4. Living with a smoker or regular exposure to secondhand smoke;
5. History of alcohol use disorder or substance use disorder of moderate or greater severity (endorsing 4 or more of the 12 criteria) in the last 12 months;
6. Acute suicidality;
7. Acute grief (<1 month);
8. Current or past psychosis;
9. Primary neurological disorder, including dementia, stroke, epilepsy, etc.;
10. MRI contraindication;
11. Electroconvulsive therapy or transcranial magnetic stimulation in last 2 months;
12. Current or planned psychotherapy;
13. Allergy or hypersensitivity to nicotine patches;
14. In the last 4 weeks, regular use of drugs with central cholinergic or anticholinergic properties or moderate / severe CYP2A6 inhibitors /inducers.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren D Taylor, MD,MHSc, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Psychiatric Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will include clinical, cognitive, and neuroimaging data from older depressed subjects. The final dataset will include clinical information about subject psychiatric diagnoses, psychiatric and medical history, cognitive data, and response to transdermal nicotine. We will share data via the National Database for Clinical Trials related to Mental Illness (NDCT). NDCT provides a secure platform for data-sharing allowing for communication of research data, tools, and supporting documents. As required by NDCT, we will obtain a Global Unique Identifier (GUID) for each participant. We will additionally follow NDCT requirements to certify and review data, as well as timeline requirements for data submission and data sharing. Sharing of neuroimaging data will also be facilitated by an XNAT system (xnat.org). XNAT is an open-source informatics software platform that assists in the management and archiving of imaging data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared according to policies from the NDCT and the NIMH Data Archive (NDA). Descriptive data, outcome measures and analyzed data will be shared will be shared within 4 months of when a publication is accepted. Study data will be shared through the NDCT indefinitely.
Access Criteria: The NIH will provide access to scientific investigators for research purposes. Qualified researchers who have completed a Data Use Certification and received approval from the NDA Data Access Committee (DAC) may be approved to access broadly shared data. A separate request process exists for access to data in federated sources. Additionally, the DAC and support staff at NIH have access to NDA shared data.
URL: https://nda.nih.gov

REFERENCES:
- [Background] Gandelman JA, Kang H, Antal A, Albert K, Boyd BD, Conley AC, Newhouse P, Taylor WD. Transdermal Nicotine for the Treatment of Mood and Cognitive Symptoms in Nonsmokers With Late-Life Depression. J Clin Psychiatry. 2018 Aug 28;79(5):18m12137. doi: 10.4088/JCP.18m12137. PMID 30192444
- [Background] Sutherland MT, Ray KL, Riedel MC, Yanes JA, Stein EA, Laird AR. Neurobiological impact of nicotinic acetylcholine receptor agonists: an activation likelihood estimation meta-analysis of pharmacologic neuroimaging studies. Biol Psychiatry. 2015 Nov 15;78(10):711-20. doi: 10.1016/j.biopsych.2014.12.021. Epub 2015 Jan 7. PMID 25662104
- [Background] Gandelman JA, Newhouse P, Taylor WD. Nicotine and networks: Potential for enhancement of mood and cognition in late-life depression. Neurosci Biobehav Rev. 2018 Jan;84:289-298. doi: 10.1016/j.neubiorev.2017.08.018. Epub 2017 Aug 30. PMID 28859996
- [Background] Aizenstein HJ, Butters MA, Wu M, Mazurkewicz LM, Stenger VA, Gianaros PJ, Becker JT, Reynolds CF 3rd, Carter CS. Altered functioning of the executive control circuit in late-life depression: episodic and persistent phenomena. Am J Geriatr Psychiatry. 2009 Jan;17(1):30-42. doi: 10.1097/JGP.0b013e31817b60af. PMID 19001356
- [Background] Alexopoulos GS, Hoptman MJ, Kanellopoulos D, Murphy CF, Lim KO, Gunning FM. Functional connectivity in the cognitive control network and the default mode network in late-life depression. J Affect Disord. 2012 Jun;139(1):56-65. doi: 10.1016/j.jad.2011.12.002. Epub 2012 Mar 15. PMID 22425432
- [Background] Taylor WD. Clinical practice. Depression in the elderly. N Engl J Med. 2014 Sep 25;371(13):1228-36. doi: 10.1056/NEJMcp1402180. No abstract available. PMID 25251617
- [Derived] Andrews P, Vega JN, Szymkowicz SM, Newhouse P, Tyndale R, Elson D, Kang H, Siddiqi S, Tyner EB, Mather K, Gunning FM, Taylor WD. Effects of open-label transdermal nicotine antidepressant augmentation on affective symptoms and executive function in late-life depression. J Affect Disord. 2024 Oct 1;362:416-424. doi: 10.1016/j.jad.2024.07.025. Epub 2024 Jul 14. PMID 39009312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from mental health clinic and the community at Vanderbilt University Medical Center in Nashville, Tennessee. Recruitment began in December, 2020 and ended in June 2022. Of 34 consented, 30 individuals met entry criteria. One participant withdrew consent prior to randomization, resulting in a final randomized sample of 29 individuals.
Pre-assignment Details: Eligible participants were only excluded for the study if they withdrew consent or for concerns for MRI safety.
Groups:
- Transdermal Nicotine Patch: Participants will wear open label transdermal nicotine patch daily for 12-15 weeks. They will apply study patch each morning and remove at bedtime. Dosage will begin at 3.5mg patch / day, increasing to a possible maximum of 21mg patch / day.
  Transdermal Nicotine patch: Participants will begin a 12- week open label trial of transdermal nicotine patch during the day and remove it at night (16 hours). Dose titration starting at 3.5 mg patch/daily to maximum of 21mg patch/daily.
  After week 12 , dose will be slowly tapered over 3 weeks.
Period: Overall Study
Arm/Group | Transdermal Nicotine Patch
Started | 29
Completed | 28
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 26
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29
Mini-Mental State Exam (MMSE) Score [Mean (Standard Deviation); unit: units on a scale] — Scale is a cognitive screening instrument. It ranges from 0-30, with higher scores indicating better cognitive performance.
  units on a scale | 29.1 (0.7)
Montgomery-Asberg Depression Rating Scale (MADRS) Score [Mean (Standard Deviation); unit: units on a scale] — This is a depression rating scale to assess depression severity. The scale ranges from 0-60, with higher scores indicating greater depression severity.
  units on a scale | 23.8 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: MADRS (Montgomery Asberg Depression Rating Scale) Score Change
Description: Primary mood outcome measured by the total score of the clinician rated MADRS. MADRS will be measured every 3 weeks (baseline, week 3, week 6, week 9, and week 12). MADRS total score range is 0-60, where higher scores indicate greater depression severity. Change is calculated as the difference between week 12 and baseline.
Time Frame: Baseline to week 12
Population: Includes 29 participants randomized, 28 of whom completed all 12 weeks and 1 completed through week 6.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
units on a scale | -15.4 (6.7)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p < 0.001, Mixed Models Analysis; Adjusted for age and gender; Slope = -1.22, Standard Error of Mean 0.12

2. Primary Outcome: Number of Participants Exhibiting Reduction in Frontal Activation During the Emotional Stroop Task During Functional Magnetic Resonance Imaging (MRI)
Description: MRI scans will be performed at baseline, week 6 and week 12. MRI will measure cognitive control network function, operationalized as a reduction in the emotional Stroop task functional MRI response in the middle and superior frontal gyri. The Stroop functional MRI response is calculated as the activation difference between incongruent and congruent conditions of the emotional Stroop task.
  The primary outcome is change in activation difference across the three time points. This is examined as a categorical variable, operationalized as those subjects who exhibit a middle / superior frontal gyri z-score reduction in activation over time of 0.5 or greater, relative to baseline at either week 6 and/or week 12. The a priori threshold being tested was that 60% or more of participants would exhibit a z-score reduction of 0.5 or greater, examined separately in the left and right middle and superior frontal gyri.
Time Frame: Baseline, week 6, week 12
Population: Includes 29 participants randomized, 28 of whom completed all 12 weeks and 1 completed through week 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 29
Participants
  Left Middle Frontal Gyrus, total region | 18
  Left Superior Frontal Gyrus, Total region | 16
  Right Middle Frontal Gyrus, total region | 17
  Right Superior Frontal Gyrus, total region | 10

3. Secondary Outcome: NIH EXAMINER Test Battery Executive Composite Score Change
Description: Secondary Cognitive Outcome: This neuropsychological test battery assesses a range of executive functions. Its Executive Composite Score is a single score that represents overall executive function performance across multiple individual neuropsychological tests, including the Dot counting test, the N-back test, the Flanker task, a continuous performance test, anti-saccades test, a set shifting test, and fluency tests. Higher scores indicate better executive function, with a range of -3.0 to 3.0. This composite is generated separately from EXAMINER sub scales.
Time Frame: Baseline to week 12
Population: Analyses includes 28 randomized participants as 1 participant withdrew at week 6 so did not complete end of study assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
units on a scale | 0.16 (0.31)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.0127, Regression, Linear; Adjusted for age, sex, education, and baseline task performance; Intercept = 0.18, 95% CI 2-sided [0.04 to 0.32], Standard Error of Mean 0.07

4. Secondary Outcome: NIH EXAMINER Test Battery Cognitive Control Factor Change
Description: Secondary Cognitive Outcome: This neuropsychological test battery assesses a range of executive functions. Its Cognitive Control Factor Score is a single score that represents cognitive control function performance across multiple individual neuropsychological tests, including the Flanker task, a continuous performance test, anti-saccades test, and a set shifting test. Higher scores indicate better executive function, with a range of -3.0 to 3.0. This is calculated independently of the executive composite or other factor scores.
  Secondary Cognitive Outcome: This neuropsychological test battery assesses a range of executive functions. We will examine its Executive Composite Score and the three factor scores (Cognitive Control, Fluency, and Working Memory). Higher scores indicate better performance.
Time Frame: Baseline to week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
units on a scale | 0.29 (0.50)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.0005, Regression, Linear; Adjusted for age, sex, education, and baseline task performance; Intercept = 0.34, 95% CI 2-sided [0.17 to 0.51], Standard Error of Mean 0.08

5. Secondary Outcome: NIH EXAMINER Test Battery Fluency Factor Change
Description: Secondary Cognitive Outcome: This neuropsychological test battery assesses a range of executive functions. Its Fluency Factor Score is a single score that represents verbal fluency performance across phonemic and categorical fluency assessments. Higher scores indicate better executive function, with a range of -3.0 to 3.0. This is calculated independently of the executive composite or other factor scores.
Time Frame: Baseline to week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
units on a scale | 0.18 (0.52)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.1027, Regression, Linear; Adjusted for age, sex, education, and baseline task performance; Intercept = 0.19, 95% CI 2-sided [-0.04 to 0.42], Standard Error of Mean 0.11

6. Secondary Outcome: NIH EXAMINER Test Battery Working Memory Factor Change
Description: Secondary Cognitive Outcome: The EXAMINER test battery Working Memory Factor Score is a single score that represents working memory performance across multiple individual neuropsychological tests, including the Dot counting and n-back tests. Higher scores indicate better executive function, with a range of -3.0 to 3.0. This is calculated independently of the executive composite or other factor scores.
  Secondary Cognitive Outcome: This neuropsychological test battery assesses a range of executive functions. We will examine its Executive Composite Score and the three factor scores (Cognitive Control, Fluency, and Working Memory). Higher scores indicate better performance.
Time Frame: Baseline to week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
units on a scale | 0.05 (0.69)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.4846, Regression, Linear; Adjusted for age, sex, education, and baseline task performance; Intercept = 0.09, 95% CI 2-sided [-0.18 to 0.37], Standard Error of Mean 0.13

7. Secondary Outcome: Choice Reaction Time (CRT) Performance Change
Description: Secondary cognitive outcome, a neuropsychological test measure of attention. We will examine change in total reaction time for the CRT. Lower reaction time indicates better performance.
Time Frame: Baseline to week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
Milliseconds | -0.67 (123.40)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.7290, Regression, Linear; Adjusted for age, sex, education, and baseline task performance; Intercept = 9.04, 95% CI 2-sided [-44.28 to 62.36], Standard Error of Mean 25.77

8. Secondary Outcome: Selective Reminding Task Performance Change
Description: Secondary cognitive outcome, Selective Reminding Task as a test of immediate and delayed verbal memory. This is an 8-trial, 16-word test where the interviewer reads unrelated words to the participant who must recall them. Any missed items are then repeated before the next attempt. Scores range from 0-60, with higher scores indicating better performance. Change in the recall over 12 weeks reflect the verbal memory function, with higher scores indicating better verbal memory performance.
Time Frame: Baseline to week12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
units on a scale | 0.33 (16.61)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.9196, Regression, Linear; Adjusted for age, sex, education, and baseline task performance; Intercept = -0.25, 95% CI 2-sided [-5.28 to 4.78], Standard Error of Mean 2.43

9. Secondary Outcome: Trait Adjectives Task, Change in Positive Items Endorsed
Description: Participants view a series of randomized, rapidly presented positive and negative characteristics and quickly indicate whether each adjective does or does not apply to them. Positive and negative adjectives are balanced. Measures include number of adjectives endorsed or rejected, and RT for those trials. These are assessed separately for positive items endorsed and negative items rejected. Task performance assesses self-referential negativity bias and is associated with antidepressant response. Task completed at baseline, week 6, and week 12. Scores for positive items endorsed range from 0 to 24, with higher scores indicating more positive items being endorsed, so a reduction in negativity bias.
Time Frame: Assessed at baseline, week 6, and week 12, change from baseline to week 12 reported
Population: Analyses includes 29 randomized participant, however 1 participant withdrew at week 6 so did not complete 12 week assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
units on a scale | 2.28 (5.55)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.033, Mixed Models Analysis; Adjusted for age and gender; Slope = 0.17, 95% CI 2-sided [0.01 to 0.33], Standard Error of Mean 0.08

10. Secondary Outcome: Trait Adjectives Task, Change in Negative Items Rejected
Description: Participants view a series of randomized, rapidly presented positive and negative characteristics and quickly indicate whether each adjective does or does not apply to them. Positive and negative adjectives are balanced. Measures include number of adjectives endorsed or rejected, and RT for those trials. These are assessed separately for positive items endorsed and negative items rejected. Task performance assesses self-referential negativity bias and is associated with antidepressant response. Task completed at baseline, week 6, and week 12. Scores for negative items rejected range from 0 to 24, with higher scores indicating that more negative items are rejected, thus a reduction in negativity bias.
Time Frame: Assessed at baseline, week 6, and week 12, change from baseline to week 12 reported
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
units on a scale | 1.92 (4.87)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.041, Mixed Models Analysis; Adjusted for age and gender; Slope = 0.18, 95% CI 2-sided [0.01 to 0.35], Standard Error of Mean 0.09

11. Secondary Outcome: Trait Adjectives Task, Change in Reaction Time to Endorse Positive Items
Description: Participants view a series of randomized, rapidly presented positive and negative characteristics and quickly indicate whether each adjective does or does not apply to them. Positive and negative adjectives are balanced. Measures include number of adjectives endorsed or rejected, and RT for those trials. These are assessed separately for positive items endorsed and negative items rejected. Task performance assesses self-referential negativity bias and is associated with antidepressant response. Task completed at baseline, week 6, and week 12. A score reduction represents increased reaction time.
Time Frame: Assessed at baseline, week 6, and week 12, change from baseline to week 12 reported
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
milliseconds | -120.99 (228.89)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.001, Mixed Models Analysis; Adjusted for age and gender; Slope = -11.13, 95% CI 2-sided [-17.81 to -4.45], Standard Error of Mean 3.36

12. Secondary Outcome: Trait Adjectives Task, Change in Reaction Time to Reject Negative Items
Description: Participants view a series of randomized, rapidly presented positive and negative characteristics and quickly indicate whether each adjective does or does not apply to them. Positive and negative adjectives are balanced. Measures include number of adjectives endorsed or rejected, and RT for those trials. These are assessed separately for positive items endorsed and negative items rejected. Task performance assesses self-referential negativity bias and is associated with antidepressant response. Task completed at baseline, week 6, and week 12. A reduction in score indicates a faster reaction time.
Time Frame: Assessed at baseline, week 6, and week 12, change from baseline to week 12 reported
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
milliseconds | -149.20 (252.25)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.001, Mixed Models Analysis; Adjusted for age and gender; Slope = -12.64, 95% CI 2-sided [-19.94 to -5.33], Standard Error of Mean 3.68

13. Secondary Outcome: Ruminative Response Scale Score Change
Description: Secondary mood outcome: Change in rumination measured by the Ruminative Response Scale total score measured at Screening visit, week 6 and week 12. This is a self-report scale with a range of 0-66, where higher scores indicate higher levels of rumination
Time Frame: Assessed at baseline, week 6, and week 12; only change in baseline to week 12 reported.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
score on a scale | -7.32 (12.27)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p < 0.001, Mixed Models Analysis; Slope = -0.74, 95% CI 2-sided [-1.15 to -0.32], Standard Error of Mean 0.20

14. Secondary Outcome: Apathy Evaluation Scale (AES) Score Change
Description: Secondary Mood Outcomes: Change in apathy as measured by the self-report AES, a questionnaire with a range of 0-54, where higher scores indicate greater apathy. Measured at baseline, week 6, and week 12.
Time Frame: Assessed at baseline, week 6, and week 12; only change in baseline to week 12 reported.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
score on a scale | -7.36 (8.91)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.001, Mixed Models Analysis; Adjusted for age and gender; Slope = -0.63, 95% CI 2-sided [-0.92 to -0.34], Standard Error of Mean 0.14

15. Secondary Outcome: Insomnia Severity Index Score Change
Description: Secondary Mood Outcomes: Change in the severity of insomnia measures as self-report , a questionnaire with the range of 0-21 ,where higher scores indicate increase in severity. Assessed at baseline, week 6, and week 12.
Time Frame: Assessed at baseline, week 6, and week 12; only change in baseline to week 12 reported.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
score on a scale | -4.50 (7.36)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p < 0.001, Mixed Models Analysis; Adjusted for age and gender; Slope = -0.41, 95% CI 2-sided [-0.65 to -0.18], Standard Error of Mean 0.12

16. Secondary Outcome: Penn State Worry Questionnaire (PSWQ) Score Change
Description: Secondary mood outcome: Change in anxiety and worry measured by PSWQ, a self-report questionnaire with a range of 16-80, where higher scores indicate greater anxiety and worry. Assessed at baseline, week 6, and week 12.
Time Frame: Assessed at baseline, week 6, and week 12; only change in baseline to week 12 reported.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
score on a scale | -5.07 (22.39)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.183, Mixed Models Analysis; Adjusted for age and gender; Slope = -0.47, 95% CI 2-sided [-1.17 to 0.23], Standard Error of Mean 0.35

17. Secondary Outcome: Fatigue Severity Scale Score Change
Description: Secondary outcome examining fatigue using a self-report questionnaire that ranges from 0- 56, where higher scores indicate more severe fatigue. Questionnaire administered at baseline, week 6, and week 12.
Time Frame: Assessed at baseline, week 6, and week 12; only change in baseline to week 12 reported.
Population: 29 participants analyzed, although one participant withdrew at week 6 before trial completion.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
score on a scale | -3.15 (14.0)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.170, Mixed Models Analysis; Analyses adjusted for age and gender; Slope = -0.30, 95% CI 2-sided [-0.74 to 0.13], Standard Error of Mean 0.22

18. Secondary Outcome: Dimensional Anhedonia Rating Scale (DARS) Score Change
Description: Secondary mood outcome: Change in anhedonia measured by DARS, a self-report questionnaire that ranges from 0-68, where lower scores indicate greater anhedonia. Conversely, higher scores indicate greater ability to enjoy activities. Assessed at baseline, week 6, and week 12.
Time Frame: Assessed at baseline, week 6, and week 12; only change in baseline to week 12 reported.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
score on a scale | 4.63 (10.47)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.051, Mixed Models Analysis; Analyses adjusted for age and gender; Slope = 0.40, 95% CI 2-sided [0.00 to 0.80], Standard Error of Mean 0.20

19. Secondary Outcome: General Anxiety Disorder-7 Item Scale (GAD7) Score Change
Description: Secondary Mood outcome: self-reported questionnaire to measure the severity of anxiety. Questionnaire ranges 0-24, higher scores indicates greater anxiety state. Assessed at baseline, week 6, and week 12.
Time Frame: Assessed at baseline, week 6, and week 12; only change in baseline to week 12 reported.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
score on a scale | -2.38 (3.37)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p < 0.001, Mixed Models Analysis; Analyses adjusted for age and gender; Slope = -0.22, 95% CI 2-sided [-0.33 to -0.11], Standard Error of Mean 0.06

20. Secondary Outcome: Patient Reported Outcome Measurement Information System (PROMIS) Applied Cognition Abilities Short Form Score Change
Description: Secondary Cognitive outcome:PROMIS (Patient reported outcome measurement information system) is a self-reported questionnaire to measure mental acuity, concentration, verbal and nonverbal memory, verbal fluency, and perceived changes in these cognitive functions, ranges from 0-32 , where higher scores indicate improvement. Assessed at baseline, week 6, and week 12.
Time Frame: Assessed at baseline, week 6, and week 12; only change in baseline to week 12 reported.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
score on a scale | 5.15 (8.27)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.002, Mixed Models Analysis; Analyses adjusted for age and gender; Slope = 0.43, 95% CI 2-sided [0.17 to 0.69], Standard Error of Mean 0.13

21. Secondary Outcome: Attentional Control Scale Score Change
Description: Secondary Attention outcome: The Attentional Control Scale (ACS) is a self-report questionnaire that has been developed to measure individual differences in attentional control. The scale ranges from 0-80, with higher scores indicative of better attentional control, and a positive change indicated improved attentional control. Assessed at baseline, week 6, and week 12.
Time Frame: Assessed at baseline, week 6, and week 12; only change in baseline to week 12 reported.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
score on a scale | 6.04 (9.96)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.002, Mixed Models Analysis; Analyses adjusted for age and gender; Slope = 0.52, 95% CI 2-sided [0.21 to 0.83], Standard Error of Mean 0.14

22. Secondary Outcome: Anxiety Sensitivity Index 3 (ASI-3) Score Change
Description: The ASI-3 is a self-report questionnaire assesses anxiety sensitivity, or the fear of arousal-related sensations. Specifically these derive from the belief that anxiety- or arousal-based sensations have negative consequences. This self-report scale includes 18 items with scores ranging from 0 to 72, where higher scores indicate greater anxiety sensitivity.
Time Frame: Assessed at baseline, Week 6, and Week 12; only baseline to week 12 reported.
Population: Includes 29 participants randomized, 28 of whom completed all 12 weeks and 1 completed through week 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 28
score on a scale | -4.40 (10.86)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.876, Mixed Models Analysis; Analyses adjusted for age and gender; Slope = 0.09, 95% CI 2-sided [-1.05 to 1.23], Standard Error of Mean 0.55

ADVERSE EVENTS:
Time Frame: Fifteen weeks
Arm/Group | Transdermal Nicotine Patch
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 26/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Nicotine Patch (N=29)
Fall (Injury, poisoning and procedural complications) | 1 (1) — Injurious fall, leading to hospitalization and surgery
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Transdermal Nicotine Patch (N=29)
Skin reaction (Skin and subcutaneous tissue disorders) | 13 — Dermatological reaction to patch site, characterized by pruritus and/or redness
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Increased tension and inner restlessness (Psychiatric disorders) | 3
Insomnia (Nervous system disorders) | 3
Increased dream activity (Nervous system disorders) | 3

LIMITATIONS AND CAVEATS:
Small, open-label study design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT04433767/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT04433767/ICF_002.pdf